CLINICAL TRIAL: NCT06817473
Title: Evaluation of the Feasibility and Efficacy of Computerized Anxiety Treatment in a Group Setting - RCT
Brief Title: Evaluation of the Feasibility and Efficacy of Computerized Anxiety Treatment in a Group Setting
Acronym: Group CAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004267
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Computerized Anxiety Sensitivity Treatment; Health Education Treatment

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of two treatment conditions (active CAST or control HET) and did not receive the other intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAST (Experimental): Computerized anxiety sensitivity treatment (CAST), which has been used by researchers already in many RCTs. This involves 30 minutes of psychoeducational video material delivered via computer presentation followed by 30 minutes of repeated interoceptive exposure practice exercises such as 60 seconds of breathing through a coffee straw, shaking head from side to side, and looking into a mirror.
  Interventions: Behavioral: CAST
- HET (Placebo Comparator): Developed as a 30-minute online intervention that provides education about physical health habits that can impact mental health, such as diet, exercise, and sleep. This intervention has been used in prior clinical trials to control for effects of general education, general coping techniques, and use of technology. Participants in past clinical trials have reported that HET is engaging and beneficial.
  Interventions: Behavioral: HET

INTERVENTIONS:
Behavioral: CAST — CAST is a transdiagnostic cognitive behavioral therapy (CBT)-based protocol designed to address elevated AS, particularly the amplification of cognitive stress symptoms including perceived confusion and memory problems. CAST is a fully computerized, 1-hour intervention. CAST contains video animation and audio narration throughout, as well as interactive features (e.g., brief quizzes to promote comprehension). Procedures draw heavily on standard CBT techniques; AS, a core vulnerability for anxiety and depression is targeted using these procedures. In this study, participants complete CAST as a group alongside other participants.
  Other Names: Computerized Anxiety Sensitivity Treatment
  Arms: CAST
Behavioral: HET — The HET protocol covers standard healthy lifestyle behaviors as well as broad coping strategies to address stress. HET is a fully computerized 1-hour control condition focused on increasing healthy behaviors and decreasing unhealthy behaviors. Content includes healthy eating, hydration, sleep and rest, stress management as well as other healthy lifestyle tips. HET was administered in a group format for this study.
  Other Names: Health Education Treatment; HEC; Health Education Control
  Arms: HET

SUMMARY:
* Statement of the Research Study. Participants are being invited to volunteer to take part in our research study. It is up to participants whether to choose to take part or not. There will be no penalty or loss of benefits to choosing not to take part or decide later not to take part.
* Purpose. The reason that the researchers are doing this research is to evaluate the effectiveness and feasibility of administering a computerized anxiety intervention in a setting of five or more individuals. This intervention has already been tested and shown promise with individuals, and researchers want to see if it will function in a group setting as well.
* Duration. Researchers think that taking part in our study will last approximately two hours, with an additional follow-up survey one month later to be completed at home via computer or smartphone.
* Research Activities. Participants will first be asked to complete several questionnaires dealing with your thoughts and feelings. Once these questionnaires are completed, participants will be assigned to one of two groups, with each group viewing one of two computerized presentations and completing some group exercises afterward. Once participants have completed the designated intervention, participants will then be asked to fill out surveys once again, which will complete the study appointment. One month following the appointment, participants will be sent surveys once again and will be asked to complete them at home.

Risks: The risks or discomforts to participants while taking part in this research include temporary distress or anxiety pr potentially feeling mild discomfort answering questions about your thoughts and feelings.

Benefits: As a result of taking part in this research, participants may experience improvements in mental health.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18+ and ability to use a computer or smartphone.

Exclusion Criteria:

* inability to engage in any interoceptive exercises.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Anxiety Sensitivity Index-3 | Baseline through Month 1 follow up
  18 item self-report measure indexing anxiety sensitivity (Taylor et al., 2007). Scores range from 0-72 with higher scores indicating more severe anxiety sensitivity
PROMIS Anxiety Scale 8a | Baseline through Month 1 Follow Up
  8-item self-report measure indexing overall anxiety (Pilkonis et al., 2011). Scores range from 8 to 40 with higher scores reflecting worse anxiety symptoms.
PROMIS Depression Scale 8b | Baseline through Month 1 Follow Up
  8 item self-report measure indexing depressive symptoms (Polkonis et al., 2014). Scores range from 8-40 with higher scores reflecting worse depression symptoms.
Treatment Acceptability Questionnaire | Baseline through Month 1 follow up
  7-item self-report measure used in prior studies (Short et al., 2017). Scores range from 0-21 with higher scores indicating more favorable acceptability ratings.
Treatment Engagement Questionnaire | Month 1 Follow Up
  Participants were given two items assessing how frequently they: 1) thought about CAST content in the past month; 2) engaged in interoceptive exposure practice.

SECONDARY OUTCOMES:
Intolerance of Uncertainty-12 | Baseline through Month 1 follow up
  12 item self-report measure indexing intolerance of uncertainty (Carleton et al., 2007). Scores range from 12-60 with higher scores reflecting worse intolerance of uncertainty.
Client Satisfaction Questionnaire | Baseline through Month 1 Follow Up
  A modified version of the Client Satisfaction Questionnaire (CSQ) will be administered to assess treatment acceptability. Scores range from 8-32 with higher scores reflecting more favorable acceptability ratings.
Difficulties in Emotion Regulation Scale | Baseline through Month 1 follow up
  16 item self-report measure indexing emotional dysregulation (DERS-16, Bjureberg et al., 2016). Scores range from 16 to 80 with higher scores reflecting worse emotion regulation difficulties.

OTHER OUTCOMES:
Group likingness/closeness | Baseline
  Self-report measure assessing how close group members felt with other members of their group (adapted from Byrne et al., 1971)
Berlin Numeracy Test | Baseline
  Brief measure of numerical ability (Cokely et al., 2011) with scores ranging from 0-4, higher scores indicate better numerical ability.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University Psychology Clinic, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schubert FT, Morabito DM, Schmidt NB. Examining the efficacy of the computerized anxiety sensitivity treatment in a guided, group format: A randomized controlled trial. Behav Res Ther. 2025 Aug;191:104785. doi: 10.1016/j.brat.2025.104785. Epub 2025 May 20. PMID 40435564